CLINICAL TRIAL: NCT02492984
Title: An Open-label, Single-arm, Post- Authorization Pragmatic Clinical Trial On The Safety And Efficacy Of Xyntha (Moroctocog-alfa (Af-cc), Recombinant Fviii) In Subjects With Hemophilia A In Usual Care Settings In China
Brief Title: PF-05208756, Moroctocog Alfa (AF-CC), Xyntha For Hemophilia A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1831083; 2015-005040-33 (EudraCT Number)
Record Dates: First submitted 2015-03-19; First posted 2015-07-09 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Hemophilia A
Keywords: FVIII inhibitor
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravenous infusions of Xyntha (Experimental): Enrolled subjects will be treated with intravenous infusions of Xyntha for: • On-Demand treatment, • Surgical Prophylaxis at a dose and frequency prescribed by the subject's treating physician in accordance with the Xyntha label and will be adjusted solely according to medical and therapeutic necessity.
  Interventions: Drug: Intravenous infusions of Xyntha

INTERVENTIONS:
Drug: Intravenous infusions of Xyntha — Enrolled subjects will be treated with intravenous infusions of Xyntha for: • On-Demand treatment, • Surgical Prophylaxis at a dose and frequency prescribed by the subject's treating physician in accordance with the Xyntha label and will be adjusted solely according to medical and therapeutic necessity.
  Other Names: Xyntha (Moroctocog-alfa (AF-CC)

SUMMARY:
An open-label, single-arm, post- authorization pragmatic clinical trial on the safety and efficacy of Xyntha (Moroctocog-alfa (AF-CC), Recombinant FVIII) in subjects with hemophilia A in usual care settings in China for approximately 6 months or or approximately 50 exposure days whichever occurs first

DETAILED DESCRIPTION:
The purpose of this post-approval study is to provide supplementary information relating to the use of Xyntha (Moroctocog-alfa (AF-CC), Recombinant FVIII) in Chinese subjects with hemophilia A, especially on the safety and efficacy in different populations of Chinese hemophilia A patients, in particular in pediatric patients <6 years of age, pediatric patients ≥6 to ≤12 years of age, Previously Untreated Patients (PUPs) , subjects receiving prophylaxis treatment after enrollment in the study, and severe patients (FVIII:C <1%).

ELIGIBILITY:
Inclusion Criteria:

* Male and/or Female subjects with Hemophilia A.
* Subjects/parents/legal representatives must be able to comply with registry procedures (informed consent/assent process, clinical visits, reporting of infusion and bleed data, reporting of adverse events, etc).
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative, parent(s)/legal guardian) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Presence of any other bleeding disorder in addition to hemophilia A.
* Treatment with immunomodulatory therapy (e.g., intravenous immunoglobulin, routine systemic corticosteroids, cyclosporins, anti-TNF agents) within 30 days prior to study entry or planned use for the duration of their study participation.
* Subjects with a past history of, or current factor VIII inhibitor. For laboratory-based assessments, any Bethesda inhibitor titer greater than the laboratory's normal range or ≥0.6 BU/mL.
* Subjects with known hypersensitivity to the active substance or to any of the excipients of Xyntha.
* Subjects with a known hypersensitivity to Chinese Hamster Ovary cell proteins.
* Unwilling or unable to follow the terms of the protocol.
* Any condition which may compromise the subject's ability to comply with and/or perform study-related activities or that poses a clinical contraindication to study participation (these conditions include, but are not limited to, inadequate medical history to assure study eligibility; expectation of poor compliance in provision of observations for study-related documentation), in the opinion of the Investigator.
* Participation in other studies involving investigational drug(s) (Phases 1-4) within 30 days before the current study begins and/or during study participation (exception for studies on Xyntha).
* Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- China (15):
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Department of Hematology,The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Department of Hematology,Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Blood Center of Shandong Province, Jinan, Shandong
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Blood Diseases Hospital, Chinese Academy of Medical Science (Institute of Hematology), Tianjin, Tianjin Municipality
  - Department of Hematology,The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Beijing Children's hospital, Beijing
  - The second affiliated hospital of chongqing medical university, Chongqing
  - Children's Hospital of Chongqing Medical University, Chongqing
  - Hematology Department, Nanfang Hospital, Southern Medical University, Guangzhou
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine/Hematology Department, Shanghai
  - Department of Hematology/Children's Hospital of Shanghai, Shanghai

REFERENCES:
- [Derived] Yang R, Zhao Y, Wang X, Sun J, Wu R, Jin C, Jin J, Wu D, Rendo P, Sun F, Rupon J, Huard F, Korth-Bradley JM, Xu L, Luo B, Liu YC. Safety and Efficacy of Moroctocog Alfa (AF-CC) in Chinese Patients with Hemophilia A: Results of Two Open-Label Studies. J Blood Med. 2020 Nov 25;11:439-448. doi: 10.2147/JBM.S241605. eCollection 2020. PMID 33269010
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As there were 2 participants who rolled over from the surgical prophylaxis group to the on-demand group should be counted once in total column, the total number of baseline participants was 85.
Groups:
- On-Demand Group: Participants were treated with intravenous infusions of Xyntha 500 International Unit (IU)/vial at a dose and frequency prescribed by the participant's treating physician in accordance with the China Xyntha Package Insert for approximately 6 months or approximately 50 exposure days (EDs).
- Surgical Prophylaxis Group: Participants were treated with intravenous infusions of Xyntha 500 IU/vial. The treatment duration for surgical prophylaxis was decided by the investigator depending on surgery nature and participant conditions.
Period: Overall Study
Arm/Group | On-Demand Group | Surgical Prophylaxis Group
Started | 73 | 14
Completed | 70 | 14
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: As there were 2 participants who rolled over from the surgical prophylaxis group to the on-demand group should be counted once in total column, the total number of baseline participants was 85.
Groups:
- Total: Total of all reporting groups
Arm/Group | On-Demand Group | Surgical Prophylaxis Group | Total
Number analyzed (Participants) | 73 | 14 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.2 (4.8) | 21.0 (15.0) | 9.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 72 | 14 | 86

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Factor VIII (FVIII) Inhibitors
Description: Percentage of participants with the product medically important event (MIE) (FVIII inhibitor development during the study).
Time Frame: From Day 1 up to 28 calendar days after End of Treatment (participants had received treatment for 6 months or when participants had achieved 50 exposure days [EDs] whichever occurred first).
Population: The safety analysis set was defined as all participants who received at least one dose of Xyntha during the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | On-Demand Group | Surgical Prophylaxis Group
Number analyzed (Participants) | 73 | 14
percentage of participants | 8.22 [3.08 to 17.04] | 7.14 [0.18 to 33.87]

2. Secondary Outcome: Number of Participants With All Causality Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence without regard to causality in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. An AE was considered treatment emergent if it started for the first time in a participant on or after the first day of active treatment, or the event started before the first day of active treatment but increased in severity during active treatment. AEs included both SAEs and non-serious AEs.
Time Frame: From Day 1 up to 28 calendar days after End of Treatment (participants had received treatment for 6 months or when participants had achieved 50 EDs whichever occurred first).
Population: The safety analysis set was defined as all participants who received at least one dose of Xyntha during the study.
Measure: Number; unit: participants
Arm/Group | On-Demand Group | Surgical Prophylaxis Group
Number analyzed (Participants) | 73 | 14
participants
  Participants with AEs | 65 | 10
  Participants with SAEs | 7 | 1

3. Secondary Outcome: Response Assessment of On-Demand Treatment of Bleeds
Description: The proportion of infusions (initial and subsequent for a bleed) in each response category (excellent, good, moderate, no response) was reported. Excellent: Definite pain relief and/or improvement in signs of bleeding starting within 8 hours after an infusion, with no additional infusion administered. Good: Definite pain relief and/or improvement in signs of bleeding starting within 8 hours after an infusion, with at least 1 additional infusion administered for complete resolution of the bleeding episode or definite pain relief and/or improvement in signs of bleeding starting after 8 hours following the infusion, with no additional infusion administered. Moderate: Probable or slight improvement starting after 8 hours following the infusion, with at least 1 additional infusion administered for complete resolution of the bleeding episode. No Response: No improvement at all between infusions or during the 24 hour interval following an infusion, or condition worsens.
Time Frame: From Day 1 up to participants had received treatment for 6 months or when participants had achieved 50 EDs whichever occurred first.
Population: Participants with a bleed during the study for which on-demand treatment with Xyntha was administered. The data for this outcome was not planned to be analyzed for the "surgical prophylaxis group".
Measure: Number; unit: percentage of infusions
Units Other Than Participants: infusions
Arm/Group | On-Demand Group
Number analyzed (Participants) | 73
Number analyzed (infusions) | 2568
percentage of infusions
  Excellent | 46.9
  Good | 40.0
  Moderate | 12.7
  No Response | 0.3
  Data Not Recorded | 0.1

4. Secondary Outcome: Number of Infusions Needed to Treat Each New Bleed for On-Demand Treatment
Description: The number of Xyntha infusions administered to treat a bleed was determined. This was calculated by adding the on-demand initial treatment and any on-demand follow-up infusions for the same bleed (same bleed start date/time).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | On-Demand Group
Number analyzed (Participants) | 73
infusions | 1.6 (0.94)

5. Secondary Outcome: Frequency of Xyntha Infusions to Treat Each New Bleed for On-Demand Group
Description: The number of bleeds resolved with 1, 2, 3, 4, or >4 infusions was reported for each of the categories (1, 2, 3, 4, or >4 infusions needed to treat the bleed), in which the numerator was the number of bleeds falling into each category, and the denominator was the total number of new bleeds across all participants.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: percentage of bleeds
Units Other Than Participants: bleeds
Arm/Group | On-Demand Group
Number analyzed (Participants) | 73
Number analyzed (bleeds) | 1610
percentage of bleeds
  1 Infusion | 63.0
  2 Infusions | 21.9
  3 Infusions | 8.6
  4 Infusions | 6.0
  >4 Infusions | 0.5

6. Secondary Outcome: Hemostatic Efficacy for Surgical Prophylaxis Treatment
Description: Assessment of hemostatic efficacy was determined by the investigator and/or surgeon using the 4 point Surgical Hemostasis Efficacy Rating Scale. Excellent: Achieved hemostasis comparable to that expected after similar surgery in a non hemophilic participant. Good: Prolonged time to hemostasis, with somewhat increased bleeding compared to that expected after similar surgery in a non hemophilic participant. Moderate: Obviously delayed hemostasis, but manageable with additional infusions. No Response: No hemostatic response. The percentage of observations in each hemostatic efficacy response category (excellent, good, moderate, none) was reported.
Time Frame: From day of surgery to postoperative period (at least 1-3 days post operation or until adequate wound healing for minor surgery or 4-6 days post operation or until threat resolved or adequate wound healing for major surgery)
Population: Surgical prophylaxis participants during their surgical prophylaxis period. The data for this outcome was not planned to be analyzed for the "on-demand group".
Measure: Number; unit: percentage of observations
Groups:
- Surgical Prophylaxis Group: Participants were treated with intravenous infusions of Xyntha 500 International Unit (IU)/vial. The treatment duration for surgical prophylaxis was decided by the investigator depending on surgery nature and participant conditions.
Arm/Group | Surgical Prophylaxis Group
Number analyzed (Participants) | 14
percentage of observations
  Day of Surgery: Excellent | 71.4
  Day of Surgery: Good | 28.6
  Day of Surgery: Moderate | 0
  Day of Surgery: None | 0
  Post-Operative: Excellent | 75.5
  Post-Operative: Good | 24.5
  Post-Operative: Moderate | 0
  Post-Operative: None | 0

7. Secondary Outcome: Actual Estimated Blood Loss for Surgical Prophylaxis Treatment
Description: Number of participants with blood loss in each category (Abnormal, Normal, and Absence). Blood loss during the intraoperative and the postoperative period were assessed by investigator or surgeon, which were rated as Abnormal, Normal, and Absence. Abnormal blood loss meant the blood loss was higher over the expectation for the non hemophilic participant.
Time Frame: as for outcome 6
Population: Surgical prophylaxis participants during their surgical prophylaxis period. The data for this outcome was not planned to be analyzed for the "on-demand group". Number of participants analyzed signifies participants evaluable for this outcome measure.
Measure: Number; unit: partcipants
Arm/Group | Surgical Prophylaxis Group
Number analyzed (Participants) | 13
partcipants
  Abnormal | 0
  Normal | 13
  Absence | 0

8. Secondary Outcome: Number of Participants With Transfusion Requirement for Surgical Prophylaxis Treatment
Description: Number of participants with transfusion requirement for surgical prophylaxis treatment. Transfusion requirements during the intraoperative and the postoperative period were assessed by investigator or surgeon. The number of units and types of blood products transfused were recorded if applicable.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Surgical Prophylaxis Group
Number analyzed (Participants) | 14
participants | 2

9. Secondary Outcome: Average Infusion Dose and Total Factor VIII Consumption for On-Demand Treatment and Surgical Prophylaxis Treatment
Description: The total amount (IU) infused for each Xyntha infusion recorded in the study drug infusion log case report form (CRF) was summed to calculate the total factor VIII consumption for each participant. The average infusion dose for each participant was calculated as his total factor VIII consumption (in IU) divided by the number of infusions administered. The total factor VIII consumption, divided by number of infusions, was summarized similarly to average infusion dose (IU).
Time Frame: On-Demand Group: Day 1 up to 6 months or 50 EDs whichever occurred first. Surgical Prophylaxis Group: Day of surgery to postoperative period. The duration of postoperative period is specified in previous endpoints.
Population: All participants who received at least one dose of Xyntha during the study
Measure: Mean (Standard Deviation); unit: International Unit (IU)
Arm/Group | On-Demand Group | Surgical Prophylaxis Group
Number analyzed (Participants) | 73 | 14
International Unit (IU)
  Average Infusion Dose | 674.68 (357.613) | 1245.07 (494.268)
  Total FVIII Consumption per Participant | 25211.0 (22035.35) | 39860.7 (27546.15)

10. Secondary Outcome: Percentage of Less Than Expected Therapeutic Effect (LETE) in the On-Demand Setting
Description: LETE occurred in the on-demand setting if 2 successive "No Response" ratings were recorded after 2 successive Xyntha drug infusions, respectively.The infusions must have been administered within 24 hours (less than or equal to 24 hours) of each other for treatment of the same bleeding event in the absence of confounding factors (prespecified). Therefore, LETE in the on-demand setting was based on the response to treatment of a bleeding episode (including those occurring during the surgical prophylaxis period). Note that on-demand treatments administered during the surgical prophylaxis period were also to be included.
Time Frame: From Day 1 up to participants had received treatment for 6 months or participants had achieved 50 EDs whichever occurred first.
Population: The safety analysis set was defined as all participants who received at least one dose of Xyntha during the study.
Measure: Number (95% Confidence Interval); unit: percentage of bleeding episodes
Units Other Than Participants: bleeding episodes
Arm/Group | On-Demand Group
Number analyzed (Participants) | 73
Number analyzed (bleeding episodes) | 1610
percentage of bleeding episodes | 0.06 [0.00 to 0.35]

11. Secondary Outcome: Number of Confirmed LETE in the Low Recovery Setting
Description: LETE could also be lower than expected recovery of FVIII in the opinion of the investigator following infusion of Xyntha in the absence of confounding factors. The only confounding factors for low recovery were: known presence or subsequent identification of a FVIII inhibitor; known compromised Xyntha; faulty administration of Xyntha, including inadequate dosing.
Time Frame: as for outcome 3
Population: The safety analysis set was defined as all participants who received at least one dose of Xyntha during the study.
Measure: Number; unit: LETE bleeds
Arm/Group | On-Demand Group | Surgical Prophylaxis Group
Number analyzed (Participants) | 73 | 14
LETE bleeds | 0 | 0

ADVERSE EVENTS:
Groups:
- Total: Treatment Group Description TBD
Arm/Group | On-Demand Group | Surgical Prophylaxis Group | Total
Serious Adverse Events (participants affected / at risk) | 7/73 | 1/14 | 8/85
Other Adverse Events (participants affected / at risk) | 62/73 | 9/14 | 70/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | On-Demand Group (N=73) | Surgical Prophylaxis Group (N=14) | Total (N=85)
Factor VIII inhibition (Blood and lymphatic system disorders) | 6 | 1 | 7
Gingival injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | On-Demand Group (N=73) | Surgical Prophylaxis Group (N=14) | Total (N=85)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Local swelling (General disorders) | 4 | 0 | 4
Peripheral swelling (General disorders) | 15 | 0 | 15
Pyrexia (General disorders) | 15 | 2 | 17
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 18 | 0 | 18
Tonsillitis (Infections and infestations) | 6 | 1 | 7
Upper respiratory tract infection (Infections and infestations) | 7 | 0 | 7
Contusion (Injury, poisoning and procedural complications) | 6 | 0 | 6
Fall (Injury, poisoning and procedural complications) | 9 | 0 | 9
Incision site oedema (Injury, poisoning and procedural complications) | 0 | 1 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 4 | 4
Joint injury (Injury, poisoning and procedural complications) | 5 | 0 | 5
Ligament sprain (Injury, poisoning and procedural complications) | 4 | 0 | 4
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 2 | 26
Arthropathy (Musculoskeletal and connective tissue disorders) | 4 | 0 | 4
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 4 | 0 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 34 | 3 | 37
Muscle swelling (Musculoskeletal and connective tissue disorders) | 11 | 0 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 0 | 18
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 2 | 2
Penile oedema (Reproductive system and breast disorders) | 0 | 1 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 10
Ecchymosis (Skin and subcutaneous tissue disorders) | 9 | 0 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 6 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from completion/termination at all participating sties. Investigator may not disclose previously undisclosed confidential information other than study results.